CLINICAL TRIAL: NCT04934254
Title: DEVELOPMENT of the NEWBORN SKIN ASSESSMENT ATTITUDE SCALE for NURSES
Brief Title: The NEWBORN SKIN ASSESSMENT ATTITUDE SCALE
Status: Completed | Type: Observational
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Adnan Batuhan Coskun, Res.Asst., Hasan Kalyoncu University
Other Study IDs: 2021-031
Record Dates: First submitted 2021-06-14; First posted 2021-06-22 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Skin Abnormalities; Newborn; Attitude of Health Personnel
Keywords: Newborn; Skin; Scale; Nurse; Construction
MeSH Terms: conditions — Skin Abnormalities

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Newborn Nurses
  Interventions: Other: Attitude Scale

INTERVENTIONS:
Other: Attitude Scale — 26-item related to scale will construct and apply to nurses for creating scale

SUMMARY:
The protection of the body integrity of the newborn is very important in terms of the development of physical and mental health and social health. Failure to protect the skin integrity of newborns and not paying attention to the clinical findings on the skin may cause morbidity/mortality. Attitudes of nurses can affect the evaluation of newborn skin negatively and/or positively.

It was determined as the development of an attitude scale for newborn nurses to evaluate newborn skin and examining the factors affecting their attitudes. In line with this purpose, an attitude scale for newborn nurses regarding the evaluation of newborn skin will be developed and nurses' attitude levels, sociodemographic variables that are related to attitude and cause significant difference can be determined.

DETAILED DESCRIPTION:
One of the indicators of the level of development of the countries is the newborn's life and death rates. The increase in the neonatal survival rate is primarily related to the care provided in the delivery room. Adaptation to the outside world is important because of the physiological and psychosocial changes experienced by the newborn after birth. For this reason, the adaptation process is monitored by monitoring the physiological and behavioral changes in the newborn.

The skin is an important organ that "protects the organism against environmental factors and also regulates temperature and water loss in the organism". Newborn skin begins to act as a barrier in the womb, matures gradually, and continues for up to 1 year after birth.

The immaturity of the skin of the newborn causes it to be the most open organ to external factors, and it has a very sensitive and fragile structure until it reaches the required maturity. Newborn skin can be damaged as a result of daily applications, and failure to follow up the skin regularly and unsuitable interventions for the skin cause morbidity/mortality.

Differences in skin maturation of preterm infants vary according to gestational age. The stratum corneum, the outer layer of the epidermis, continues to mature until the 24th - 34th week of pregnancy. In preterm infants born before the stratum corneum is mature; Risks of infection, transepidermal water loss, temperature irregularity, absorption of topical agents, or physical trauma are encountered.

In order for neonatal nurses to fulfill their duties and responsibilities; They should have knowledge and skills such as evaluating the newborn, using the equipment and technologies in the unit, training/counseling parents, communicating effectively and collaborating. While providing appropriate care by neonatal nurses increases the effect of the treatment, it also minimizes the side effects that may occur. It is also very important for the early diagnosis and treatment of the problems that have occurred and/or may occur with the clinical findings determined as a result of the skin evaluation of the newborn by the nurses.

Attitude is one of the processes in which the individual is involved and has an important place in explaining the reason for the behavior of the individual. Attitude is a preparatory tendency for behavior and is the result of the interaction of emotion, thought and behavior elements. The fact that the individual has order, harmony and continuity between his feelings, thoughts and behaviors regarding a situation/event shows that a positive attitude towards that situation/event is developed.

When the national and international literature on nurses, who have an important role in the evaluation of newborn skin, is examined, there are studies examining the knowledge and skills of skin evaluation and care of both healthy and risky newborns. However, nowadays, it is observed that instead of using an objective assessment tool, whose validity and reliability has been ensured, in the evaluation of the skin condition of especially healthy/risky newborns, the definitions of 'impaired skin integrity' or 'complete skin integrity' are still made with the evaluations made with a subjective approach, and the newborn skin is not considered as a whole. Regular evaluation of newborn skin is part of good care and allows for early diagnosis and treatment of skin problems. In the evaluations made with a subjective approach, the definitions of 'impaired skin integrity' or 'skin integrity' are made, and the skin is not considered as a whole.

In the national and international literature review, assumptions and opinions regarding newborn nurses' evaluation of newborn skin with a subjective approach rather than an objective approach have been put forward, but no research has been encountered that examines their attitudes towards the subject. It is known that nurses' attitudes towards evaluating newborn skin are important for the early prevention of skin problems of newborns and other problems that may develop due to these problems, as an indicator of their tendencies towards the evaluation process.

ELIGIBILITY:
Inclusion Criteria:

●After obtaining written consent and informed consent form from neonatal nurses who agreed to participate in the study, they will be included in the study.

Exclusion Criteria:

* Written permission cannot be obtained,
* Nurses who do not work with newborns,
* Participants included in the sample in the development of the attitude scale will be excluded from the study in the final form application.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The nurses who work in Newborn intensive care unit
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2021-03-30 (Actual); Primary Completion 2022-10-20 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
Scale Development Process | 3 months
  94 questions will prepare as "Nurse Opinion Determination Form for "Newborn Skin Attitude" and 16 newborn nurses' opinions will collect.
Scale creation | 1 month
  Measuring instrument consisting items will create. In order to determine the comprehensibility and content validity of the scale, it was presented to at least 20 experienced nurses
Validity and reliability of scale | 6 months
  After final agreement of scale items, it will apply to at least 300 nurses for construction and psychometric analysis

CONTACTS AND LOCATIONS:
Overall Officials: Güven Hoş, Study Director — Hasan Kalyoncu University
Locations (1):
- Hasan Kalyoncu University, Gaziantep, Şahinbey, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Fernandes JD, Machado MC, Oliveira ZN. Children and newborn skin care and prevention. An Bras Dermatol. 2011 Jan-Feb;86(1):102-10. doi: 10.1590/s0365-05962011000100014. English, Portuguese. PMID 21437530
- [Background] Suddaby EC, Barnett S, Facteau L. Skin breakdown in acute care pediatrics. Pediatr Nurs. 2005 Mar-Apr;31(2):132-8, 148. PMID 15934568
- [Background] Murdoch V. Pressure care in the paediatric intensive care unit. Nurs Stand. 2002 Oct 23;17(6):71-4, 76. PMID 12434752
- [Background] Rayner G, Blackburn J, Edward KL, Stephenson J, Ousey K. Emergency department nurse's attitudes towards patients who self-harm: A meta-analysis. Int J Ment Health Nurs. 2019 Feb;28(1):40-53. doi: 10.1111/inm.12550. Epub 2018 Nov 1. PMID 30387232
- [Background] Djaja N, Youl P, Aitken J, Janda M. Evaluation of a skin self examination attitude scale using an item response theory model approach. Health Qual Life Outcomes. 2014 Dec 24;12:189. doi: 10.1186/s12955-014-0189-x. PMID 25539671